CLINICAL TRIAL: NCT07009613
Title: Integration of Strongyloides Stercoralis Public Health Control Into the Soil-transmitted Helminths Control Programme in Rwanda - The SCAN Study
Brief Title: Strongyloides Stercoralis Public Health Control in Rwanda
Acronym: SCAN
Status: Completed | Type: Observational
Sponsor: IRCCS Sacro Cuore Don Calabria di Negrar (Other)
Collaborators: University of Rwanda (Other); Rwanda Biomedical Centre (Other)
Responsible Party: Principal Investigator, Dora Buonfrate, Head of infectious disease Clinical Research Unit, IRCCS Sacro Cuore Don Calabria di Negrar
Other Study IDs: No477/RNEC/2024
Record Dates: First submitted 2025-05-17; First posted 2025-06-06 (Actual); Last update posted 2025-06-06 (Actual); Status verified 2025-06

CONDITIONS: Strongyloides Stercoralis Infection; Strongyloides
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Parasitological tests — The primary outcome was reported based on the technicians' answers collected with a structured questionnaire. The individuals screened underwent testing with the tests detailed above
Other: Questionnaire — The primary outcome was based on the technicians' evaluation, based on their answers collected in a questionnaire. The individuals screened were tested with assays used for the national control programmes

SUMMARY:
The World Health Organization (WHO) recently issued guideline for the public health control of Strongyloides stercoralis in endemic areas. We aimed to evaluate the feasibility of implementing the WHO recommendations in Rwanda, specifically to intergrate the activities for the public health control of strongyloidiasis in the ongoing national programme for the control of the other soil-transmitted helminths and schistosomiasis, that has been in place for several years. As additional objective, we aimed to estimate the prevalence of S. stercoralis in two districts of Rwanda (Gisagara and Rubavu). To evaluate the feasibility, we asked lab technicians to evaluate challenges emerged during the implementation of the laboratory procedures with a structured questionnaire. Also, we evaluated the costs needed to perform these tests. We estimated the prevalence of S. stercoralis by calculating the number of positive cases out of all people tested. The lab technicians participated to a training session, where they were taught the S. stercoralis-specific lab techniques, and to a two-day pilot study where they could practice. The tests used were parasitological techniques (agar stool culture, (APC) and Baermann method) and an antibody rapid diagnostic test (RDT). Duration of training, with a specific focus on larvae differentiation, was identified as pivotal for a successful implementation of the parasitological techniques. The use of the RDT was instead considered easy to apply at all evaluation time points. Raw cost (i.e. not including staff salaries and transport costs) of materials and equipment was below 2 euros/test for each assay. In both districts, Strongyloides prevalence was below the threshold recommended by the WHO for the implementation of mass treatment, hence this aspect was not evaluated.

ELIGIBILITY:
Inclusion Criteria:

* People living in the selected districts and households
* Obtainment of written informed consent (for children's participation, consent was sought from parents/guardians).

Exclusion Criteria:

* Inability to supply an adequate stool sample

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes
Study Population: People living in two districts in Rwanda
Sampling Method: Probability Sample
Enrollment: 1415 (Actual)
Dates: Start 2024-09-23 (Actual); Primary Completion 2024-10-11 (Actual); Study Completion 2024-10-14 (Actual)

PRIMARY OUTCOMES:
Evaluation of the tests based on technicians' perception (through questionnaire) and costs | The data will be collected at baseline, during the pilot study (two - three days from baseline) and during field work (after two to three weeks from baseline)
  Technicians' previous experience with each S. stercoralis-specific assay, along with their perceptions regarding the ease of each of the procedural steps and associated safety concerns were assessed using a structured questionnaire. Each procedural step was rated as "Very easy", "Easy", "Neutral", "Difficult" and "Very difficult". For the steps marked "difficult" or "very difficult", respondents could specify the reasons for the difficulty from a predefined non-mutually-exclusive list of options. The per-test costs were calculated from the procurement records of each S. stercoralis-specific assay.

SECONDARY OUTCOMES:
Prevalence | through study completion
  Frequency of S. stercoralis cases out of the tested population

CONTACTS AND LOCATIONS:
Locations (1):
- School of Health Sciences, College of Medicine and Health Sciences, University of Rwanda, Kigali, Rwanda

IPD SHARING:
Plan to Share IPD: No